CLINICAL TRIAL: NCT03983070
Title: The Effects of Lower Extremity Blood Flow Restriction Training on Power, and Muscle Size.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campbell University, Incorporated (Other)
Responsible Party: Principal Investigator, Bradley Myers, Assistant Professor, Campbell University, Incorporated
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 491
Record Dates: First submitted 2019-05-31; First posted 2019-06-12 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: Strength; Hypertrophy; Oxygen consumption
MeSH Terms: conditions — Hypertrophy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with parallel groups
Who Masked: Outcomes Assessor
Masking Description: Blinded researcher will perform preliminary and outcomes measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Exercise Group (Active Comparator): Participants allocated to the Control Exercise Group will participate in 8 total exercise sessions (2x per week for 4 weeks). Exercise sessions will include two exercise modalities 1)seated rowing ergometer and 2) dumbbell deadlifts. Exercise intensity will be individualized based upon preliminary testing with rowing at 80% maximal Watts, and deadlifts at 60% of one-repetition maximum.
  Interventions: Other: Seated Rowing Ergometer; Other: Deadlift
- Blood Flow Restriction and Exercise Group (Experimental): Participants allocated to the Control Exercise Group will participate in 8 total exercise sessions (2x per week for 4 weeks). Exercise sessions will include the application of blood flow restriction during two exercise modalities 1)seated rowing ergometer and 2) dumbbell deadlifts. Exercise intensity will be individualized based upon preliminary testing with rowing at 40% maximal Watts, and deadlifts at 30% of one-repetition maximum. Blow flow restriction will be applied at 80% occlusion during both exercise modalities.
  Interventions: Other: Seated Rowing Ergometer; Other: Deadlift; Other: Blood flow restriction

INTERVENTIONS:
Other: Seated Rowing Ergometer — Seated rowing exercise performed at a specific percentage of maximal Watts according to pre-intervention measures
Other: Deadlift — Deadlift exercise performed with a set of dumbbell weights at a sepcific percentage of pre-intervention one-repetition maximum.
Other: Blood flow restriction — An occlusive cuff will be placed around each proximal thigh and inflated to 80% arterial occlusion during exercise sessions.
  Arms: Blood Flow Restriction and Exercise Group

SUMMARY:
Blood-flow restriction training (BFR) is a technique utilized to provide the benefits of high intensity exercise (strength, power, hypertrophy) when applied to exercise intensities that are insufficient to produce these benefits without BFR. The technique involves the application of an occlusive cuff (similar in design to a blood pressure cuff) over the limb of an individual that is set to occlude arterial blood flow at a given percentage during exercise. BFR has demonstrated increased strength and muscle hypertrophy compared to control interventions in various populations including: healthy subjects, athletes, post-surgery, clinical rehabilitation, and older adults.

Most research on BFR has been conducted on single joint exercises and not exercises that exhibit more complex movements typically associated with daily activities. The early evidence of complex exercises combined with BFR suggests that strength and hypertrophy both improve, however more research needs to be conducted.

The purpose of this project is to determine if four weeks of BFR training combined with approach rowing and deadlifts increases strength, power, aerobic capacity, and muscle size. These results will be compared to an isovolumetric control.

DETAILED DESCRIPTION:
INITIAL DATA COLLECTION (60-75 minutes) Measurements will be performed by a researcher blinded to group allocation. Height and weight will be measured with a stadiometer and calibrated scale.

Participant will sit to complete the following intake forms: Par-Q+, Numeric Pain Rating Scale, International Physical Activity Questionnaire- short form After sitting at least 5 minutes the following resting measures will be taken: resting heart rate, resting blood pressure

Thigh Circumference (supine): Markings will be made bilaterally at the lateral femoral condyle, proximal greater trochanter, and a line in an anterior to posterior direction 50% between these two landmarks. A circumferential measurement of the thigh will be taken three separate times at that 50% line for each leg.

Muscle Size: Measurements will be taken of the vastus lateralis and biceps femoris following the protocol established by Ruas et al using the GE LOGIC e, GE Healthcare, WI, USA). Superficial markings will be made to assist the researcher in locating desired anatomical location for measurement. Markings will be made bilaterally at the lateral femoral condyle, proximal aspect of greater trochanter, and a line in an anterior to posterior direction 50% between these two landmarks. Participants will lay supine for vastus lateralis and prone for biceps femoris measurement. The ultrasound transducer will be placed on the skin, utilizing a water-gel coupling agent, oriented perpendicular to the skin interface over the muscle of interest at the line that marks 50% of the distance between lateral femoral condyle and proximal greater trochanter. Images will be saved in the ultrasound device using participant identifier, muscle visualized, and date (example: BFR01_VL_05.01.19). Images will be exported to a computer for analysis using ImageJ software (National Institutes of Health, Bethesda, MD, USA).

Maximal Vo2: Oxygen consumption will be assessed on stationary rower (Concept2 Inc., Morrisville, VT) utilizing a metabolic cart and gas exchange (ParvoMedics, Provo, UT). Throughout the exercise test rating of perceived exertion (RPE) will be assessed within the final 10 seconds of each stage. Each participant will proceed throughout the various stages of the exercise test in a sequential fashion until test is terminated for one of the following reasons (1) participant requests to stop exercise test, (2) RPE reaches 10 out of 10, (3) participant fails to maintain desired Watts for that stage.

Maximal Deadlift Test:

Lower extremity strength will be assessed through an estimated one-repetition maximum (1-RM) deadlift with a dumbbell in each hand. Prior to performing the test each participant will receive instruction on proper technique for deadlift and the ability to perform practice repetitions as needed. The participant will begin with an estimated weight after consultation with research team member. The participant will grasp one dumbbell in each hand in an upright standing position and perform the maximum number of deadlifts possible. If the participant performs at least 1 repetition and no more than 9 repetitions of deadlifts they are finished with the deadlift test. If the participant performs more than 9 repetitions the resistance will be altered following the table below and the deadlift test will be performed again after 2-minute rest. Periods of testing and rest will alternate until the resistance provides at least 1 repetition but no more than 9 repetitions. The final deadlift weight and number of successful repetitions will be recorded and entered into the following equation to determine an estimated maximum deadlift resistance.

Randomization Participants will be randomly assigned to either the BFR group or the control group (CG), using block randomization. A predetermined random allocation of equal parts BFR and CG will be determined for each set of 10 participants (example: participants 1-10 will contain a random allocation of 5 to each intervention group, the same for participants 11-20 and 21-30). The block randomization will be performed by an individual not involved in this study (other than to randomize) with the result of the randomization being concealed until the after initial testing session. Both groups will participate in the same number of exercise sessions (2x per week for 4 weeks) and one final testing session.

EXERCISE SESSIONS (Study total = 4 hours) All exercise sessions will be conducted by a researcher who is not blinded to group allocation. Each group will complete two training sessions per week for four weeks. RPE will be recorded in the final seconds of each round of exercise. If participant does not complete the protocol for either rower or deadlift the resistance will be retained for future sessions. If participant reports <6/10 RPE at the final stage of either rower or deadlift the intensity for that exercise will be increased by 10% (watts or resistance respectively).

BFR Group

BFR will be conducted utilizing the Personal Tourniquet System (PTS) for BFR, Delfi Medical Innovations Inc (Vancouver , BC, Canada).

WARM-UP: Standard dynamic warm-up

BFR Set-up

1. Placement of BFR sleeve and BFR cuffs around bilateral thighs.
2. Participant will lay supine with cuffs in place.
3. Researcher will initiate cuff inflation to measure arterial pressure
4. After successful measurement of arterial pressure each cuff will be set to inflate to 80% occlusion for the exercise session.
5. Participant will remain in BFR cuffs and move into the exercise session. Participants will complete a dynamic warm-up prior to starting the BFR exercise protocol. Upon completion of the protocol, the cuff will be deflated and removed. The participant will then walk for five minutes at a self-selected pace for a cool down.

Control Group

Participants will complete an identical dynamic warm-up as the BFR group prior to starting the CG exercise protocol. Upon completion of the protocol, the participant will then walk for five minutes at a self-selected pace for a cool down.

Final Testing Protocol (60-75 minutes)

Follow the same protocol as initial testing with all measurements taken by researcher blinded to group allocation. The researcher conducting final testing will not have been involved in the intervention period for any participant nor ask the participant about their experience or group allocation. Participants will also be instructed to not share their group allocation with the researcher collecting the final data.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active adults (3 mo more days of moderate intensity physical activity per week, with at least some combination of aerobic and strength training).

Exclusion Criteria:

* Failure to achieve clearance for exercise participation via the Par-Q+ screening tool
* Currently pregnant or with 3 months post-partum
* Presence of chronic low back pain
* history of surgery to change the structure of joints within the lower extremity (joint replacement, osteotomy)
* Known blood clotting disorder or taking blood thinner medications
* Presence of peripheral vascular disease
* Presence of systemic or widespread pain disorder (fibromyalgia, chronic regional pain syndrome)
* Currently under activity limitations for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Size after 4 weeks | after 4 weeks of intervention
  Cross-sectional measurement of muscle girth

SECONDARY OUTCOMES:
Change in Maximal Oxygen Consumption after 4 weeks | after 4 weeks of intervention
  Oxygen consumption will be assessed utilizing a metabolic cart and gas exchange during maximal effort seated rowing ergometry.
Change in Maximal Deadlift Strength after 4 weeks | after 4 weeks of intervention
  One-repetition maximum strength will be assessed through incremental mass increases and estimation once participant can lift no more than 9 repetitions.

OTHER OUTCOMES:
Change in Numeric Pain Rating after 4 weeks | after 4 weeks of intervention
  Numeric Pain Rating Scale (0-10). Participants will rate their present experience of pain from 0 "no pain" to 10 "worst imaginable pain." Participants can select any whole number, higher scores represent more intense pain experience. This scale contains only one verbal question.
Change in International Physical Activity Questionnaire - Short Form after 4 weeks | after 4 weeks of intervention
  Assessment of physical activity over 7 day period
Change in Resting Heart Rate after 4 weeks | after 4 weeks of intervention
  After 5 minutes of seated rest heart rate will be assessed
Change in Resting Blood Pressure after 4 weeks | after 4 weeks of intervention
  After 5 minutes of seated rest blood pressure will be assessed
Chang in Thigh circumference after 4 weeks | after 4 weeks of intervention
  Cicumferential measures of the thigh 50% of the way between greater trochanter and lateral femoral condyle

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J Myers, DPT, DSc, Principal Investigator — Campbell University
Locations (1):
- Campbell University, Buies Creek, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No